CLINICAL TRIAL: NCT06740617
Title: Evaluation Of Balance And Ankle Proprioception In Calcaneal Spur Patients
Acronym: CS
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Afifi Saad Mohamed Farahat, principle investigator: mai afifi saad farahat, Cairo University
Other Study IDs: P.T.REC/012/005501
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Calcaneal Spur
Keywords: calcaneal spur; balance; ankle proprioception
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- calcaneal spur group: twenty six patients with calcaneal spur will participate in this group
- healthy group: twenty six healthy subjects will participate in this group

SUMMARY:
this study will be conducted to investigate the difference in balance and ankle proprioception between calcaneus spur patients and age matched normal subjects

DETAILED DESCRIPTION:
A calcaneal spur, also known as enthesophyte, is an abnormal bone outgrowth at the inferior part of the calcaneus, which is the most common site of bony spur occurrence. Although there is consensus that a calcaneal spur is a common cause of heel pain, approximately 20% of calcaneal spurs are asymptomatic and its pathology remains not fully understood.Ankle Joint Position Sense (JPS) refers to the ability to accurately perceive and reproduce the position of the ankle joint in space. Balance, on the other hand, encompasses the ankle joint's positional stability during both static and dynamic activities.Several investigations have demonstrated a significant association between ankle JPS and balance, indicating that individuals with better proprioceptive acuity in the ankle joint tend to exhibit superior postural stability, ). It was found that higher plantar fascia and heel fat pad stiffness and thickness are related to higher postural sway in anterior-posterior and medial-lateral directions based on the single-leg balance tests. These results suggest that the morphological and mechanical properties of plantar fascia and heel fat pad play an important role in balance performance.

ELIGIBILITY:
Inclusion Criteria:

* age will range from 40-60
* both sex male and female
* unilateral calcaneal spur
* Patients with pain and inflammation at the bottom of heel, or the location where the spur is present.
* All subjects have body mass index less than 29 kg/cm2
* sharp pain like a knife in the heel when standing up in the morning
* pain may also appear at the end of the day or after spending long periods of time on the feet
* sharp pain with the first steps in the morning or after a long period of rest and dissipating when weight bearing is initiated.
* All diagnosed patients, were evaluated and confirmed radiologically by specialist doctor, by performing a standard X-ray foot profile image

Exclusion Criteria:

* Surgery within the last 6 months
* Sensory or motor paralysis -Received steroid injections within the last 3 months-
* discrepancy in length of the lower extremities greater than or equal to 1 cm.
* systemic disease in the last six months that may predispose to heel pain(e.g., rheumatoid arthritis and lupus). (Dudoniene V et al.,2023).
* Calcaneal spurs are associated with various medical conditions, including obesity, rheumatoid arthritis, osteoarthritis, ankylosing spondylitis, Reiter's disease, and spondylarthritis.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: fifty two subjects will be assigned to two group; group with calcaneal spur and healthy group
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
dynamic balance | up to one day
  the Biodex Balance System (BBS) ,Version 3.1, has been used to evaluate postural balance
static balance | up to one day
  The single-leg stance balance test will be used to assess static balance.
ankle propriception | up to one day
  digital inclinometer will be used to assessed ankle proprioception
foot disability | up to one day
  A Foot Function Index (FFI) will be used to assess foot disability. The pain subcategory consists of 9 items and measures foot pain in different situations, such as walking barefoot versus walking with shoes. The disability subcategory consists of 9 items and measures difficulty performing various functional activities because of foot problems, such as difficulty climbing stairs. The activity limitation subcategory consists of 5 items and measures limitations in activities because of foot problems, such as staying in bed all day. Recorded on a visual analogue scale (VAS), scores range from 0 to 100 mm, with higher scores indicating worse pain. Both total and subcategory scores are calculated

SECONDARY OUTCOMES:
integrity of the plantar fascia ligament | up to one day
  The Windlass Test is a physical examination technique will be used to assess the integrity of the plantar fascia ligament in the foot. we evaluated the Windlass test, and found it had a high specificity, and a low level of sensitivity. It can be used as part of the clinician's armamentarium in evaluating patients with plantar fasciitis, and should be performed in a weightbearing position to maximize the sensitivity